CLINICAL TRIAL: NCT03574740
Title: Influence of Tobacco Smoking on the Development of Obstructive Sleep Apnea (OSA)
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, Principal Investigator, Astes
Other Study IDs: Tobacco-OSA
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Obstructive Sleep Apnea; Tobacco Use
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tobacco Use | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Entire population: All patients included in this retrospective study. These patients were analyzed following their tobacco smoking habits.
  Interventions: Other: Tobacco Smoking

INTERVENTIONS:
Other: Tobacco Smoking — Influence of Tobacco Smoking on the development of OSA

SUMMARY:
The aim of this study was to retrospectively evaluate the influence of Tobacco Smoking on the development of Obstructive Sleep Apnea (OSA).

DETAILED DESCRIPTION:
The aim of this study was to retrospectively evaluate the influence of Tobacco Smoking on the development of Obstructive Sleep Apnea (OSA).

Statistical analysis will be performed on this retrospective population to determine in tobacco smoking could influence the development of OSA.

ELIGIBILITY:
Inclusion Criteria:

* All patients for a preoperative anesthetic consultation between 01/01/14 and 31/12/17 who undergo a polysomnography

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for a preoperative anesthetic consultation between 01/01/14 and 31/12/17 who undergo a polysomnography. For these patients, the influence of tobacco smoking on the development of OSA will be studied.
Sampling Method: Probability Sample
Enrollment: 1298 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Obstructive Sleep Apnea (OSA) | 1 month
  Diagnosis of OSA based on a polysomnography recording

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, PhD, Principal Investigator — Astes

IPD SHARING:
Plan to Share IPD: No